CLINICAL TRIAL: NCT06554730
Title: Non-interventional Post-authorization Study of Belzutifan in Adult Patients With Von Hippel-Lindau Disease-associated Renal Cell Carcinoma, Pancreatic Neuroendocrine Tumor and/or Central Nervous System Hemangioblastoma (MK-6482-026)
Brief Title: MSD Belzutifan PAS
Status: Withdrawn | Type: Observational
Why Stopped: Study is registered /active on RWD Catalogues (https://catalogues.ema.europa.eu) - Please refer to EU PAS number: EUPAS108114
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-0221; MK-6482-026 (Other: MSD Belzutifan); NCI-2024-06807 (Registry Identifier: Clinical Trials Reporting Program); EUPAS108114 (Registry Identifier: RWD Catalogues - EU PAS)
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Von Hippel Lindau Disease
Keywords: Belzutifan; VHL
MeSH Terms: conditions — von Hippel-Lindau Disease | interventions — belzutifan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — This study has been registered and will be maintained through close out on the RWD Catalogues Observational Registry - https://catalogues.ema.europa.eu/ under the EU PAS number: EUPAS108114
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Belzutifan — There is no intervention for this study. This study will be collecting data from the EMR of consenting subjects who are taking Belzutifan.

SUMMARY:
This is a prospective observational cohort study evaluating the effectiveness and safety of belzutifan treatment in routine clinical practice.

This study has been registered and will be maintained through close out on the RWD Catalogues Observational Registry - https://catalogues.ema.europa.eu/ under the EU PAS number:

EUPAS108114

DETAILED DESCRIPTION:
Primary Objective

* Among new users of belzutifan with VHL disease-associated RCC, to describe the proportion of patients who undergo at least one renal tumor reductive surgery (e.g., nephrectomy) or locally directed therapy (e.g., radiofrequency ablation).
* Among new users of belzutifan with VHL disease-associated CNS hemangioblastoma, to describe the proportion of patients who undergo at least one CNS tumor reductive surgery (e.g., craniectomy) or locally directed therapy (e.g., radiation therapy).

Secondary Objectives

Among all new users of belzutifan to describe:

- Proportion of patients with treatment emergent SAEs, including the nature of these events.

Treatment patterns including the:

* Duration of therapy
* Proportion of patients who discontinued treatment, time to treatment discontinuation, and summary of reasons for discontinuation
* Proportion of patients who interrupted treatment, time to treatment interruption, duration of treatment interruption, and summary of reasons for treatment interruption
* Proportion of patients with dose reductions, and reason for dose reduction.
* Among new users of belzutifan with VHL disease-associated RCC and, separately, VHL disease-associated CNS hemangioblastoma, to describe:
* Proportion of patients who develop metastatic disease (for RCC only)
* Proportion of patients with occurrence of new VHL disease-associated tumor or tumor type

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Diagnosed with VHL disease based on a germline test or clinical diagnosis
* A decision has been made by the treating physician (at his/her discrestion) to intitate the first belzutifan treatment (i.e., belzutifan 'new users'), within the prescribing conditions of the approved product label
* Signed informed consent prior to or withing 30 days after the first inititaion of belzutifan

Exclusion Criteria:

* Anti-cancer systemic therapy within 2 weeks prior to the index date
* Unable to consent to participate in the study
* History of VHL disease-related metastasis or advanced cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedure | Through study completion
  Proportion of patients who undergo surgery or other tumor reductive procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- See also: HMA-EMA Catalogues of real-world data: EU PAS number: EUPAS108114 — https://catalogues.ema.europa.eu/node/3892/administrative-details